CLINICAL TRIAL: NCT07044908
Title: A Phase Ib/II Clinical Study Evaluating TQB2922 for Injection and Chemotherapy in Combination With or Without Bevacizumab in Subjects With RAS/BRAF Wild-Type Advanced Colorectal Cancer Who Have Failed Chemotherapy
Brief Title: TQB2922 and TAS-102 Tablets for Injection With or Without Bevacizumab in Chemotherapy-failed RAS/BRAF Wild-type Advanced Colorectal Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TQB2922-Ib/II-01
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-04

CONDITIONS: RAS/BRAF Wild Type Colorectal Cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TQB2922 injection + TAS-102 tablets (Experimental): Phase Ib: TQB2922 injection + TAS-102 tablets; TQB2922 is administered in the appropriate dose group, intravenously, every 28 days, once weekly in cycle 1 and every 2 weeks starting in cycle 2; TAS-102 tablets are administered at 35 mg/m2 (maximum 80 mg in a single dose), orally, twice daily, repeated every 28 days, on days 1 to 5 and 8 to 12. The dosage will be repeated every 28 days.
  Interventions: Drug: TQB2922 injection ± TAS-102 tablets
- TQB2922 injection (Experimental): Phase Ib: TQB2922 injection; TQB2922 is administered in the appropriate dose group, intravenously, every 28 days, once weekly in cycle 1 and every 2 weeks starting in cycle 2; TAS-102 tablets are administered at 35 mg/m2 (maximum 80 mg in a single dose), orally, twice daily, repeated every 28 days, on days 1 to 5 and 8 to 12. The dosage will be repeated every 28 days.
  Interventions: Drug: TQB2922 injection ± TAS-102 tablets
- TQB2922 injection+TAS-102 tablets + Bevacizumab (Experimental): Phase II: TQB2922 injection + TAS-102 tablets + bevacizumab; TQB2922 will be administered according to Recommended Phase 2 Dose (RP2D), one treatment cycle every 28 days, and once a week in the first cycle.
  TQB2922 was administered according to RP2D, one treatment cycle every 28 days, once a week in the 1st cycle, and once every 2 weeks starting from the 2nd cycle; TAS-102 tablets were administered at 35 mg/m2 (maximum 80 mg in a single dose) orally twice a day on days 1-5 and 8-12, and repeated every 28 days; bevacizumab was administered at 5 mg/kg intravenously on the 1st day, and repeated every 2 weeks.
  Interventions: Drug: TQB2922 injection+TAS-102 tablets ± Bevacizumab
- TQB2922 injection+TAS-102 tablets (Experimental): Phase II: TQB2922 injection + TAS-102 tablets; TQB2922 will be administered according to RP2D, one treatment cycle every 28 days, and once a week in the first cycle.
  TQB2922 was administered according to RP2D, one treatment cycle every 28 days, once a week in the 1st cycle, and once every 2 weeks starting from the 2nd cycle; TAS-102 tablets were administered at 35 mg/m2 (maximum 80 mg in a single dose) orally twice a day on days 1-5 and 8-12, and repeated every 28 days; bevacizumab was administered at 5 mg/kg intravenously on the 1st day, and repeated every 2 weeks.
  Interventions: Drug: TQB2922 injection+TAS-102 tablets ± Bevacizumab

INTERVENTIONS:
Drug: TQB2922 injection ± TAS-102 tablets — TQB2922 is an anti-EGFR/c-Met bispecific antibody, subtype Immunoglobulin G1 (IgG1). TQB2922 blocks the activation of EGFR and c-Met signalling pathway by binding to EGFR and c-Met on the surface of tumour cells, thus preventing tumour growth and progression. At the same time, TQB2922 can target EGFR and c-Met on the surface of tumour cells through antibody-dependent cytotoxicity (ADCC) and antibody-dependent cell phagocytosis by natural killer cells and macrophages, thus killing tumour cells.
  Arms: TQB2922 injection; TQB2922 injection + TAS-102 tablets
Drug: TQB2922 injection+TAS-102 tablets ± Bevacizumab — TQB2922 is an anti-EGFR/c-Met bispecific antibody, subtype IgG1. TQB2922 blocks the activation of EGFR and c-Met signalling pathway by binding to EGFR and c-Met on the surface of tumour cells, thus preventing tumour growth and progression. At the same time, TQB2922 can target EGFR and c-Met on the surface of tumour cells through antibody-dependent cytotoxicity (ADCC) and antibody-dependent cell phagocytosis by natural killer cells and macrophages, thus killing tumour cells.
  Arms: TQB2922 injection+TAS-102 tablets; TQB2922 injection+TAS-102 tablets + Bevacizumab

SUMMARY:
This is a multicenter, open Phase Ib/II clinical study evaluating the safety and efficacy of TQB2922 in combination with TAS-102±bevacizumab in subjects with RAS/BRAF wild-type unresectable locally advanced or metastatic colorectal cancer that has failed treatment with oxaliplatin, fluorouracil-based and irinotecan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily enrolled in the study, signed the informed consent and had good compliance;
* Age: 18-75 years old (including boundaries at the time of signing the informed consent);
* Eastern Cooperative Oncology Group (ECOG) score: 0-1;
* Expected survival of more than 3 months;
* Unresectable locally advanced or metastatic colorectal cancer diagnosed by histological/cytological pathology;
* Disease progression or intolerable after prior treatment with oxaliplatin, fluorouracil-based and irinotecan and treated with cetuximab or bevacizumab;
* Patients with genetic testing showing wild-type for both rat sarcoma (RAS) and B-type rapid response protein kinase (BRAF);
* Presence of at least 1 measurable lesion according to RECIST 1.1 criteria;
* Laboratory tests meet the criteria;
* Female subjects of childbearing potential must agree to use contraception (e.g., Intrauterine Device (IUD), birth control pills, or condoms) for the duration of the study and for 6 months after the end of the study; must have a negative serum pregnancy/urine pregnancy test
* within 7 days prior to study entry and must not be breastfeeding; male subjects must agree to use contraception for the duration of the study and for 6 months after the end of the study.

Exclusion Criteria:

* Patients who have had previous confirmation of microsatellite high instability/mismatch repair defects (MSI-H/dMMR) by immunohistochemistry (IHC), next-generation sequencing (NGS) or polymerase chain reaction (PCR);
* Presence of a disease that interferes with intravenous administration, intravenous blood collection, or multiple factors that interfere with oral administration of medications (e.g., inability to swallow, chronic diarrhoea and intestinal obstruction);
* Active inflammatory bowel disease (ulcerative colitis, Crohn's disease) within 28 days prior to first dose;
* The presence or current concurrent presence of other malignancies within 2 years prior to the first dose.
* Unresolved toxic reactions above Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 due to any prior therapy, excluding alopecia, fatigue and peripheral neuropathy;
* Major surgical treatment, incisional biopsy or significant traumatic injury within 28 days prior to first dose;
* The presence of a long-standing unhealed wound or fracture;
* Cerebrovascular accident (including temporary ischaemic attack, cerebral haemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism within 6 months prior to the first dose;
* Have a history of psychotropic substance abuse and are unable to quit or have a mental disorder;
* Subjects with any severe and/or uncontrolled medical condition, including:

  * Unsatisfactory control of blood pressure (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg, at least 2 measurements taken at intervals of more than 24h);
  * Myocardial infarction, unstable angina pectoris, stable angina pectoris ≥ Grade 2, heart failure ≥ Grade 2 (New York Heart Association (NYHA) classification), arrhythmia ≥ Grade 2;
  * Active or uncontrolled severe bacterial, viral, or systemic fungal infection (≥ CTC AE grade 2 infection) within 28 days prior to first dose; patients with active tuberculosis within 1 year prior to enrolment.
  * Active viral hepatitis with poor control. Subjects will be screened if they meet the following requirements: Hepatitis B surface antigen (HBsAg) positive subjects with Hepatitis B virus (HBV) DNA quantification <2000 IU/ml (or 1*10 4 copy/ml) or at least 1 week of anti-HBV treatment with a 10-fold (1 log) or greater reduction in viral index prior to study entry. Subject is willing to remain on anti-HBV therapy for the entire duration of the study; HCV-infected patients (HCV Ab or HCV RNA positive) who are judged to be stable by the investigator or who are on antiviral therapy at the time of enrolment and who continue to receive approved antiviral therapy during the study;
  * Subjects with a history of (non-infectious) interstitial lung disease requiring systemic steroid therapy, or current interstitial lung disease/interstitial pneumonia; or subjects with Screening Imaging suggestive of suspected interstitial lung disease/interstitial pneumonia that cannot be ruled out;
  * History of immunodeficiency, including being human immunodeficiency virus (HIV) positive or having other acquired, congenital immunodeficiency diseases;
  * Poorly controlled diabetes mellitus (fasting blood glucose (FBG) > 10 mmol/L); and
  * Active syphilis infection.
* Known tumour-associated spinal cord compression, cancerous meningitis, with symptoms of brain metastases, or symptoms controlled for less than 4 weeks;
* Imaging suggestive of tumour invasion of large blood vessels or, in the judgement of the investigator, there is a high probability of tumour rupture or invasion of vital blood vessels during the study period leading to fatal haemorrhage;
* Failure to control a plasma (thoracic, abdominal, or pericardial) effusion that requires repeated drainage;
* Local radiotherapy within 2 weeks or >30% bone marrow irradiation radiotherapy for bone metastases within 4 weeks prior to first dose.
* Chemotherapy, targeted therapy, immunotherapy, or other antineoplastic agents within 4 weeks prior to the first dose, or who are still on drug 5.

treatment, or subjects who are still within 5 half-lives of the drug (whichever occurs first);

* Prior use of epidermal growth factor receptor/c-mesenchymal epidermal transforming factor (EGFR/c-Met) dual-antibody drugs;
* Received treatment with a proprietary Chinese medicine with an anti-tumour indication as specified in the National Drug
* Administration (NMPA) approved drug insert within 1 week prior to study treatment.
* History of live attenuated vaccination within 2 weeks prior to the first dose or planned live attenuated vaccination during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Baseline up to 48 weeks
  One or more unacceptable toxic reactions following administration of the drug, resulting in the inability to continue increasing the dose or prolonging the dosing cycle.
Objective Response Rate (ORR) | Complete response time was achieved, evaluation is expected to take 1 years.
  Proportion of patients with tumour volume reduction to a pre-specified value that maintains the minimum timeframe requirement.

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 48 weeks
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD.
Incidence of adverse event (AE) and serious adverse event (SAE) | Baseline up to 48 weeks
  The incidence and severity of adverse events were determined according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 rating scale
Disease Control Rate (DCR) | Complete response time was achieved, evaluation is expected to take 1 years.
  The proportion of subjects who achieved complete response (CR), partial response (PR), or stable disease (SD) was assessed.
Recommended Phase 2 Dose | Baseline up to 48 weeks
  The dose recommended for Phase 2 trials based on Phase 1 safety, tolerability, and pharmacokinetic data.
Elimination Half-life | Baseline up to 48 weeks
  The time required for the plasma concentration of a drug to decrease by 50% during the elimination phase, reflecting metabolic and excretory rates.
Area Under the Curve | Baseline up to 48 weeks
  The integral of the drug concentration-time curve in plasma, representing total systemic drug exposure.
Apparent Clearance | Baseline up to 48 weeks
  The apparent volume of plasma cleared of the drug per unit time, typically expressed in L/h.
Apparent Volume of Distribution in Terminal Phase | Baseline up to 48 weeks
  The apparent volume in which a drug is distributed during the terminal phase, calculated based on plasma concentration, indicating tissue distribution extent.
Trough Concentration | Baseline up to 48 weeks
  The plasma drug concentration measured at the end of a dosing interval (before next administration), used to assess accumulation risk.
Duration of Response | Complete response time was achieved, evaluation is expected to take 1 years.
  Time from first documented objective response (e.g., tumor shrinkage) to disease progression or death.
Progression-Free Survival | 1 year of assessment is expected from the start of enrolment to the first occurrence of disease progression or death from any cause
  Time from enrollment to disease progression or death from any cause, evaluating treatment's disease control ability.
Incidence of Anti-Drug Antibody | Baseline up to 48 weeks
  The proportion of patients developing antidrug antibodies during treatment, indicating immunogenicity risk.

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - National Cancer Center/Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Shantou University Medical College Affiliated Cancer Hospital, Shantou, Guangdong
  - Guangxi Zhuang Autonomous Region Cancer Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Xinyang Central Hospital, Xinyang, Henan
  - Zhoukou Central Hospital, Zhoukou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Suzhou Municipal Hospital, Suzhou, Jiangsu
  - Jiangnan University Affiliated Hospital, Wuxi, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Yibin First People's Hospital, Yibin, Sichuan